CLINICAL TRIAL: NCT02231697
Title: The RECENSUS Study: A Medical Chart Review of Patients With X-Linked Myotubular Myopathy (XLMTM)
Brief Title: A Medical Chart Review of Patients With X-Linked Myotubular Myopathy (XLMTM)
Status: Completed | Type: Observational
Sponsor: Astellas Gene Therapies (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: ATX-MTM-001 RECENSUS
Record Dates: First submitted 2014-08-28; First posted 2014-09-04 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Males With X-linked Myotubular Myopathy (XLMTM)
Keywords: XLMTM
MeSH Terms: conditions — Myopathies, Structural, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- XLMTM patients - deceased: Non-interventional, retrospective medical chart review
  Interventions: Other: Non-interventional, retrospective medical chart review
- XLMTM patients - living: Non-interventional, retrospective medical chart review
  Interventions: Other: Non-interventional, retrospective medical chart review

INTERVENTIONS:
Other: Non-interventional, retrospective medical chart review — Non-interventional, retrospective medical chart review

SUMMARY:
This retrospective medical chart review (RECENSUS) of approximately 100 XLMTM patients (with a goal to obtain 50 deceased and 20 living records) will provide further knowledge about the clinical manifestations and recorded medical management of XLMTM and potentially inform the design of future therapeutic intervention studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with XLMTM resulting from a confirmed mutation in the MTM1 gene, or a combination of XLMTM genetically confirmed family history and muscle biopsy
* Patient is male
* Access to available medical records for each patient
* Signed informed consent by the parent(s) or legal guardians and/or assent by the patient (when applicable), unless the associated IRB provides an appropriate consent waiver

Exclusion Criteria:

* Patient data after participation in an interventional study designed to treat XLMTM (patient data prior to participation in an interventional study may be included)

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Males with X-linked myotubular myopathy
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2014-09; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Survival | Lifetime, up to 50 years
  Descriptive statistics: mean, median, range for age at death for deceased patients, mean, median, range for current age for living patients

SECONDARY OUTCOMES:
Age at diagnosis | Lifetime, up to 50 years
  Descriptive statistics: mean, median, range for age of definitive diagnosis
Age at tracheostomy (if applicable) | Lifetime, up to 50 years
  Descriptive statistics: mean, median, range for number of patients requiring tracheostomy (if applicable) and average age at tracheostomy
Age at need for/type of ventilation (if applicable) | Lifetime, up to 50 years
  Descriptive statistics: mean, median, range for number of patients requiring ventilation (if applicable) and type of ventilation

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Cure CMD, San Pedro, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Florida - Gainesville, Children's Research Institute, Gainesville, Florida
  - Lurie Children's Hospital, Chicago, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - Royal Manchester Children's Hospital, Manchester

REFERENCES:
- [Derived] Graham RJ, Muntoni F, Hughes I, Yum SW, Kuntz NL, Yang ML, Byrne BJ, Prasad S, Alvarez R, Genetti CA, Haselkorn T, James ES, LaRusso LB, Noursalehi M, Rico S, Beggs AH. Mortality and respiratory support in X-linked myotubular myopathy: a RECENSUS retrospective analysis. Arch Dis Child. 2020 Apr;105(4):332-338. doi: 10.1136/archdischild-2019-317910. Epub 2019 Sep 4. PMID 31484632